CLINICAL TRIAL: NCT00378599
Title: PROTECT - Pegylated Interferon Alfa-2b and Ribavirin After Orthotopic Liver Transplantation: Efficacy and Safety in Hepatitis C Recurrence Therapy
Brief Title: Effects of Pegylated Interferon Alfa-2b and Ribavirin After Orthotopic Liver Transplantation in Subjects With Chronic Hepatitis C Recurrence (P04590AM3)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04590
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Results first posted 2010-07-16 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: Liver Transplantation; Hepatitis C, Chronic; Liver Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Liver Cirrhosis | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PEG-Intron plus Rebetol (RBV) (Experimental): PEG-Intron plus RBV treatment for up to 48 weeks with 24-week follow up. SCH 54031 PEG-Intron 1.5 ug/kg SC per week plus SCH 18908 REBETOL twice daily (BID) PO with food, dosed as followed: Weeks 1 and 2, RBV Dose 400 mg (2 capsules, 1 AM and 1 PM). At the end of Weeks 2 and 4 of Treatment (tx), a complete blood count (CBC) was performed. An increase in RBV dose was permitted only if the hemoglobin was >10 g/dL. At Weeks 3 and 4, RBV dose was 800 mg (4 capsules, 2 AM and 2 PM). From Weeks 5 to 48, RBV doses could be increased based on subject body weight. For subjects weighing <65 kg, maximum dose of RBV was to be 800 mg (4 capsules, 2 AM and 2 PM), for subjects weighing 65-85 kg, max dose of RBV was 1000 mg/day (5 capsules, 2 AM and 3 PM), for subjects weighing >85 kg, max dose of RBV was 1200 mg/day, 6 capsules, 3 AM and 3 PM).
  Interventions: Drug: Combination of (a) pegylated interferon alfa-2b and (b) rebetol

INTERVENTIONS:
Drug: Combination of (a) pegylated interferon alfa-2b and (b) rebetol — 1. Powder for injection in vials and Redipen (50, 80, 120, and 150 microgram strengths), subcutaneous, dose of 1.5 micrograms/kg, weekly for up to 48 weeks
  2. 200 mg capsules, oral, weight based dose of 400-1200 mg, daily for up to 48 weeks
  Other Names: (a) SCH 54031, PEG-Intron; (b) SCH 18908, Rebetol

SUMMARY:
This is an exploratory study and is a Phase 3, single-arm, multi-center, open-label study of pegylated interferon alfa-2b, PEG-IFN alpha-2b (PEG-Intron) and ribavirin (RBV) to determine the sustained virologic response (SVR) at 24-week follow-up to 48 week in subjects after orthotopic liver transplantation (OLT) with chronic hepatitis C (HCV) recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must confirm that all prior medication washout times have been observed.
* Subject must be 18 - 70 years of age of either gender and of any race.
* Subject must be transplanted for end-stage hepatitis C or fulminant hepatitis C.
* Subject must have documented:

  * persistent HCV viremia after OLT as defined by plasma positive for HCV RNA by quantitative reverse transcription-polymerase chain reaction (RT-PCR),
  * A liver transplant performed at least 3 months prior to screening but not more than 3 years prior to screening.
* Subject must be on stable doses of immunosuppression for at least 1 month.
* Compensated liver disease with minimum hematologic, biochemical, and serologic criteria at the (Day 1) baseline visit.

  * Alpha-fetoprotein value (AFP) less than or equal to 250ng/mL. If AFP greater than 100 ng/mL, patient will need evidence of normal liver (magnetic resonance imaging) MRI and normal chest computerized tomography (CT) scan within the last 3 months or during the screening period.
* For subjects with a history of diabetes or hypertension, clearance from an ophthalmologist has to be obtained prior to treatment start (Day 1/Visit 2).
* Subjects with a history of mild depression may be considered for entry into this study.
* Female subjects cannot be pregnant or breastfeeding and must be either postmenopausal, surgically sterile or using 2 methods of birth control.
* Sexually active male subjects are practicing an acceptable, method of contraception.
* Contraceptive measures will be reviewed with female subjects at each visit. Dual methods of contraception must be used for 1 month prior to the start of treatment and 6 months after treatment discontinuation.
* Pregnancy tests obtained at Screen Visit and Day 1 Visit prior to the initiation of treatment must be negative.

Exclusion Criteria:

* Pregnant women, women who plan to become pregnant, male subjects whose partner wants to become pregnant, and breastfeeding women (during study and up to 6 months after study completion).
* Subject has used any investigational product within 30 days prior to Screening or is participating in any other clinical study.
* Prior treatment for chronic hepatitis C post-liver transplant, including but not limited to antiviral or immunomodulatory product, any interferon product, or RBV, either as monotherapy or in combination.
* Subjects with other organ transplants.
* Any subject who received a positive hepatitis C core antibody (HBcAb) or HCV positive donor liver graft.
* Retransplantation of the liver for rejection or graft failure.
* Evidence of decompensated liver disease.
* Known coagulopathies including hemophilia.
* Known hemoglobinopathies.
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency.
* Hypersensitivity to alpha interferon and/or RBV.
* Co-infection with hepatitis B virus (HBV) and/or human immunodeficiency virus (HIV).
* Evidence of active or suspected malignancy or a history of malignancy within the last 5 years (with the exception of pre-transplant hepatocellular carcinoma histologically within the Milan criteria, and adequately treated basal or squamous cell carcinoma of the skin).
* Any known pre-existing medical condition that could interfere with the subject's participation in and completion of the study.
* Subject is or was a substance abuser. Subjects treated with buprenorphine (Subutex) who have been stable for 6 months may be included.
* Patients weighing over 135 kg;

Is participating in any other clinical study(ies);

Is allergic to or has sensitivity to the study drug or its excipients.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gordon FD, Kwo P, Ghalib R, Crippin J, Vargas HE, Brown KA, Schiano T, Chaudhri E, Pedicone LD, Brown RS Jr. Peginterferon-alpha-2b and ribavirin for hepatitis C recurrence postorthotopic liver transplantation. J Clin Gastroenterol. 2012 Sep;46(8):700-8. doi: 10.1097/MCG.0b013e31825833be. PMID 22739223

RESULTS

PARTICIPANT FLOW:
Groups:
- PEG-Intron Plus Ribavirin: PEG-Intron plus ribavirin treatment for up to 48 weeks with 24-week follow up
Period: Overall Study
Arm/Group | PEG-Intron Plus Ribavirin
Started | 125
Completed | 73
Not Completed | 52
Not completed — Adverse Event | 38
Not completed — Protocol Violation | 2
Not completed — Treatment failure | 7
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | PEG-Intron Plus Ribavirin
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 106

OUTCOME MEASURES:

1. Primary Outcome: A Sustained Virologic Response (SVR), Defined as a Plasma HCV RNA Level Below the Lower Level of Quantitation (LLQ) at 24 Weeks Post-treatment
Description: Number of participants with SVR at 24-week follow up after treatment with PEG-Intron and Ribavirin in post-orthotopic liver transplant recipients with recurrent HCV.
Time Frame: 24 weeks after completion of up to 48 weeks of therapy
Population: Intent to Treat (ITT) Data Set: All enrolled subjects who received at least one dose of any study medication (PEG-Intron or Rebetol (RBV)). Analysis of all primary and secondary efficacy endpoints and safety variables was based on the ITT population.
Measure: Number; unit: Participants
Arm/Group | PEG-Intron Plus Ribavirin
Number analyzed (Participants) | 125
Participants | 36 [21.1 to 37.6]
Statistical Analysis 1: Comparison: PEG-Intron Plus Ribavirin; Test type: Superiority or Other; Binomial Approximation = .288, 95% CI 2-sided [0.21 to 0.38]

ADVERSE EVENTS:
Arm/Group | Pegylated Interferon Alfa-2b and Ribavirin
Serious Adverse Events (participants affected / at risk) | 32/125
Other Adverse Events (participants affected / at risk) | 125/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon Alfa-2b and Ribavirin (N=125)
ANAEMIA (Blood and lymphatic system disorders) | 5 (5)
LEUKOPENIA (Blood and lymphatic system disorders) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 2 (4)
NAUSEA (Gastrointestinal disorders) | 2 (3)
VOMITING (Gastrointestinal disorders) | 3 (4)
ASTHENIA (General disorders) | 1 (1)
CHEST PAIN (General disorders) | 3 (3)
CHILLS (General disorders) | 1 (1)
MALAISE (General disorders) | 2 (2)
PYREXIA (General disorders) | 2 (2)
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 1 (1)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1)
LIVER TRANSPLANT REJECTION (Immune system disorders) | 2 (3)
APPENDICITIS (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 3 (3)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 (2)
GASTROENTERITIS (Infections and infestations) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1)
OSTEOMYELITIS (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 4 (4)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
ANASTOMOTIC COMPLICATION (Injury, poisoning and procedural complications) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1)
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 3 (3)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 3 (3)
SYNCOPE (Nervous system disorders) | 1 (1)
DRUG ABUSE (Psychiatric disorders) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
TREATMENT NONCOMPLIANCE (Social circumstances) | 1 (1)
LEG AMPUTATION (Surgical and medical procedures) | 1 (1)
SPLENECTOMY (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegylated Interferon Alfa-2b and Ribavirin (N=125)
ANAEMIA (Blood and lymphatic system disorders) | 91 (162)
LEUKOPENIA (Blood and lymphatic system disorders) | 17 (25)
NEUTROPENIA (Blood and lymphatic system disorders) | 39 (51)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 16 (20)
VISION BLURRED (Eye disorders) | 11 (11)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 12 (13)
ABDOMINAL PAIN (Gastrointestinal disorders) | 13 (19)
CONSTIPATION (Gastrointestinal disorders) | 8 (9)
DIARRHOEA (Gastrointestinal disorders) | 51 (73)
DRY MOUTH (Gastrointestinal disorders) | 11 (11)
NAUSEA (Gastrointestinal disorders) | 59 (72)
STOMATITIS (Gastrointestinal disorders) | 15 (15)
VOMITING (Gastrointestinal disorders) | 32 (44)
ASTHENIA (General disorders) | 10 (13)
CHILLS (General disorders) | 28 (28)
FATIGUE (General disorders) | 89 (112)
INFLUENZA LIKE ILLNESS (General disorders) | 18 (22)
INJECTION SITE ERYTHEMA (General disorders) | 16 (17)
INJECTION SITE RASH (General disorders) | 7 (7)
IRRITABILITY (General disorders) | 27 (27)
MALAISE (General disorders) | 7 (11)
OEDEMA PERIPHERAL (General disorders) | 9 (10)
PAIN (General disorders) | 18 (20)
PYREXIA (General disorders) | 35 (49)
INFLUENZA (Infections and infestations) | 8 (8)
SINUSITIS (Infections and infestations) | 7 (9)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 (8)
BLOOD CREATININE INCREASED (Investigations) | 10 (13)
WEIGHT DECREASED (Investigations) | 29 (30)
ANOREXIA (Metabolism and nutrition disorders) | 15 (16)
DECREASED APPETITE (Metabolism and nutrition disorders) | 33 (38)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 8 (9)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 26 (29)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 20 (22)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 11 (13)
MYALGIA (Musculoskeletal and connective tissue disorders) | 21 (22)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 (11)
DIZZINESS (Nervous system disorders) | 31 (36)
HEADACHE (Nervous system disorders) | 79 (98)
HYPOAESTHESIA (Nervous system disorders) | 8 (10)
TREMOR (Nervous system disorders) | 7 (7)
ANXIETY (Psychiatric disorders) | 19 (21)
DEPRESSION (Psychiatric disorders) | 29 (36)
INSOMNIA (Psychiatric disorders) | 39 (41)
COUGH (Respiratory, thoracic and mediastinal disorders) | 18 (23)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 32 (37)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 15 (17)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 12 (14)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 7 (7)
ALOPECIA (Skin and subcutaneous tissue disorders) | 13 (13)
DRY SKIN (Skin and subcutaneous tissue disorders) | 12 (12)
PRURITUS (Skin and subcutaneous tissue disorders) | 18 (19)
RASH (Skin and subcutaneous tissue disorders) | 32 (41)
HYPERTENSION (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Lead investigator agrees not to publish or publicly present any interim results of the Study without prior written consent of the sponsor. Lead investigator further agrees to provide 45 days written notice to the sponsor prior to submission for publication or presentation to permit the sponsor to review copies of abstracts or manuscripts for publication, which report any results of the Study. Sponsor shall have the right to review and comment on any presentation, including editorial rights.